CLINICAL TRIAL: NCT01011179
Title: An Internet-based Self-management Program With Telephone Support for Adolescents With Arthritis: A Pilot Randomized Controlled Trial
Brief Title: Internet Self-Management Program With Telephone Support for Adolescents With Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Arthritis Patient Alliance (Other); Provincial Health Services Authority British Columbia (Other); Dalhousie University (Other); IWK Health Centre (Other); The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000010809
Record Dates: First submitted 2009-09-28; First posted 2009-11-11 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Teens Taking Charge; Managing Arthritis Online; juvenile idiopathic arthritis; internet; self-management
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based JIA Self-Management Program (Experimental)
  Interventions: Behavioral: Teens Taking Charge
- Attention Control Group (Active Comparator)
  Interventions: Behavioral: Self-Management

INTERVENTIONS:
Behavioral: Teens Taking Charge — The intervention is a 12-week multi-component treatment protocol that consists of self-management strategies (e.g., how to deal with stress and treatment related symptoms like pain), information (e.g., common problems associated with treatment and disease) and social support (e.g., monitored discussion boards and narratives in the form of written stories and video clips). It will be delivered on a restricted web-site and through regular contact with a trained coach by means of email and/or telephone using standardized scripts.
  Arms: Internet-based JIA Self-Management Program
Behavioral: Self-Management — Adolescents' "own best efforts" at managing their JIA
  Arms: Attention Control Group

SUMMARY:
This study will evaluate the feasibility of "Teens Taking Charge: Managing Arthritis On-line" intervention that will help adolescents with arthritis to better manage their disease and improve their health-related quality of life (HRQL).

DETAILED DESCRIPTION:
This feasibility study will (1) assess adolescents' willingness to be randomized; (2) pilot the intervention, attention control strategies (e.g., adolescents' 'own best efforts' at managing arthritis), and outcome measures; (3) determine adolescents' perceptions regarding acceptability of the web-based intervention; and (4) obtain estimates of treatment effects in primary (HRQL) and secondary (knowledge, coping, self-efficacy, stress, treatment adherence, pain) outcome measures to inform the calculation of appropriate sample size for the future RCT.

We hypothesize that adolescents with JIA in the web-based intervention will demonstrate: (a) improved HRQL; (b) increased disease-specific knowledge; (c) improved coping, self-efficacy, and adherence to prescribed management; and (d) decreased pain and stress compared to adolescents in the attention control group

ELIGIBILITY:
Inclusion Criteria:

* adolescents 12 to 18 years
* diagnosed with JIA,
* able to speak and read English or French
* able to complete baseline online outcome measures.

Exclusion Criteria:

* cognitive impairment
* major co-morbid illnesses (medical or psychiatric) which may impact their ability to understand and use the web-based program.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, MD, Principal Investigator — IWK Health Centre
Locations (4):
- Canada (4):
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Center, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec

REFERENCES:
- [Result] Stinson JN, McGrath PJ, Hodnett ED, Feldman BM, Duffy CM, Huber AM, Tucker LB, Hetherington CR, Tse SM, Spiegel LR, Campillo S, Gill NK, White ME. An internet-based self-management program with telephone support for adolescents with arthritis: a pilot randomized controlled trial. J Rheumatol. 2010 Sep;37(9):1944-52. doi: 10.3899/jrheum.091327. Epub 2010 Jul 1. PMID 20595280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 pediatric, rheumatology clinics located within tertiary care centers across Canada. Adolescent participants were recruited between October and November 2008.
Groups:
- Attention Control Group: Self-Management : Adolescents' "own best efforts" at managing their JIA
- Internet-based JIA Self-Management Program: Teens Taking Charge : The intervention is a 12-week multi-component treatment protocol that consists of self-management strategies (e.g., how to deal with stress and treatment related symptoms like pain), information (e.g., common problems associated with treatment and disease) and social support (e.g., monitored discussion boards and narratives in the form of written stories and video clips). It will be delivered on a restricted web-site and through regular contact with a trained coach by means of email and/or telephone using standardized scripts.
Period: Overall Study
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program
Started | 24 | 22
Completed | 20 | 20
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 22 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Juvenile Arthritis Quality of Life Questionnaire (JAQQ)
Description: The questionnaire is divided into 4 dimensions: gross motor function, fine motor function, psychosocial function, and general symptoms. A 7-point ordinal scale is used to rate responses to each item from 1 (none of the time) to 7 (all of the time), based on how often the item was a problem for the child over the past 2 weeks. Total score was composed of the 4 dimension scores (top 5 items of that dimension) divided by 4, with higher scores denoting poorer HRQOL.
Time Frame: Baseline (prior to randomization) and 3 months after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet-based JIA Self-Management Program | Attention Control Group
Number analyzed (Participants) | 22 | 24
units on a scale
  Baseline | 2.35 (1.34) | 2.74 (1.36)
  Post-intervention | 1.95 (1.40) | 2.27 (1.21)

2. Secondary Outcome: Medical Issues Sub-Scale From Medical Issues, Exercise, Pain, and Social Support Questionnaire (MEPS)
Description: Measure looks at disease specific knowledge. Subscale used: Medical Issues Subscale scores range from 0 (min) - 10 (max) with higher scores indicating greater knowledge.
Time Frame: 3 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program
Number analyzed (Participants) | 24 | 22
score on a scale | 4.16 (1.96) | 6.98 (1.08)

3. Secondary Outcome: Pain Coping (Pain Coping Questionnaire)
Time Frame: Baseline (prior to randomization) and 3 months after intervention
Population: Data was not collected for this measure
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Children's Arthritis Self-Efficacy Scale (CASE)
Description: Measure looks at Self-efficacy. Subscales: Activity, Emotion, Family. Subscale scores range 0 - 10 with higher scores indicating greater self-efficacy.
Time Frame: 3 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program
Number analyzed (Participants) | 24 | 22
score on a scale
  Symptom Standard Score | 6.55 (2.75) | 7.47 (1.89)
  Emotional Standard Score | 8.11 (2.22) | 7.96 (2.38)
  Activity Standard Score | 7.60 (2.72) | 7.88 (2.42)

5. Secondary Outcome: Child Adherence Report Questionnaire (CARQ)
Description: Measure examines adherence to treatment. Subscales: Treatment Adherence to: Medication, Exercise, Splints. Subscale scores rage 0 - 10 with higher scores indicate better overall child ability in relation to following treatment recommendations.
Time Frame: 3 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program
Number analyzed (Participants) | 24 | 22
score on a scale
  Medication | 7.5 (2.96) | 8.14 (8.14)
  Exercise | 4.68 (3.26) | 5.05 (3.78)

6. Secondary Outcome: Perceived Stress Questionnaire (PSQ)
Description: Measure examines stress. Total score calculated was an average of all items with a range from 1-4 with higher scores indicating greater stress.
Time Frame: 3 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program
Number analyzed (Participants) | 24 | 22
score on a scale | 2.13 (0.42) | 1.98 (0.42)

ADVERSE EVENTS:
Arm/Group | Attention Control Group | Internet-based JIA Self-Management Program
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No